CLINICAL TRIAL: NCT03674294
Title: Efficacy of Aprepitant for the Prevention of Chemotherapy-induced Nausea and Vomiting in Nondrinking Women Younger Than 50 Years Who Received Moderately Emetogenic Chemotherapy: A Randomized, Double-blind, Phase Ⅲ Trial
Brief Title: Aprepitant Triple Therapy for the Prevention of CINV in Nondrinking and Young Women Who Received Moderately Emetogenic Chemotherapy
Acronym: CINV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yuhong Li, Director, Department of Medical Oncology, Principal Investigator, Clinical Professor, Yuhong Li, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Aprepitant-CINV
Record Dates: First submitted 2018-04-18; First posted 2018-09-17 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Gastrointestinal Neoplasms; Chemotherapy-induced Nausea and Vomiting
MeSH Terms: conditions — Gastrointestinal Neoplasms; Vomiting | interventions — Aprepitant; Palonosetron; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Palonosetron/Dexamethasone/Aprepitant (Experimental)
  Interventions: Drug: Aprepitant; Drug: Palonosetron; Drug: Dexamethasone
- Palonosetron/Dexamethasone/Placebo (Placebo Comparator)
  Interventions: Drug: Palonosetron; Drug: Dexamethasone; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Aprepitant — Aprepitant is manufactured by Merck & Co. for prevention of acute and delayed chemotherapy-induced nausea and vomiting (CINV) and for prevention of postoperative nausea and vomiting. It was approved by the FDA in 2003
  Arms: Palonosetron/Dexamethasone/Aprepitant
Drug: Palonosetron — Palonosetron is a 5-HT3 antagonist used in the prevention and treatment of chemotherapy-induced nausea and vomiting (CINV). It is used for the control of delayed CINV-nausea and vomiting and there are tentative data to suggest that it may be more effective than granisetron.
Drug: Dexamethasone — Dexamethasone is a type of corticosteroid medication. It is used in the treatment of many conditions, including rheumatic problems, a number of skin diseases, severe allergies, asthma, chronic obstructive lung disease, croup, brain swelling, and along with antibiotics in tuberculosis.
Drug: Placebo Oral Tablet — In the current clinical trial, placebo oral tablet is provided as a substance for Aprepitant with no active therapeutic effect.
  Arms: Palonosetron/Dexamethasone/Placebo

SUMMARY:
The purpose of this study is to study whether adding Aprepitant to Palonosetron and dexamethasone can further prevent the incidence and severity of nausea and vomiting caused by FOLFIRI or FOLFOX chemotherapy regimen among gastrointestinal malignancy patients with high risk factors of chemotherapy-associated adverse events.

DETAILED DESCRIPTION:
The purpose of this study is to study whether adding Aprepitant to Palonosetron and dexamethasone can further prevent the incidence and severity of nausea and vomiting caused by FOLFIRI or FOLFOX chemotherapy regimen after curative effect among gastrointestinal malignancy patients with high risk factors of chemotherapy-associated adverse events.This study will observe and evaluate the incidence and severity of nausea and vomiting as well as the effectiveness of corresponding treatment(with or without Aprepitant) during Day 1 to Day 5 from the beginning of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed by pathology as gastrointestinal carcinoma and no previous FOLFOX or FOLFIRI based regimen chemotherapy history.
* Female.
* Adult patients ( ≥ 18, ≤ 50 years of age)
* No long-term or excessive alcohol intake history:1.Alcohol intake less than 5 times per week; 2.Alcohol intake less than 100g per day.
* Performance status ECOG 0-1
* Adequate haematological, hepatic, renal and metabolic function parameters:

Leukocytes : 3,500-10,000/mm3, ANC ≥ 1,500/mm3, Platelets ≥ 90,000/mm3, Hb > 9g/dl (may be transfused or treated with erythropoietin to maintain or exceed this level), Serum creatinine ≤ 1 x upper limit of normal, Bilirubin ≤ 1.5 x upper limit of normal, Serum AST, ALT, ALP ≤ 2.5 x upper limit of normal in absence of liver metastases, or ≤ 5 x upper limit of normal in presence of liver metastases.

* Negative pregnancy test. If pregnancy test were positive, subject should be included in the trial only when the subsequent pregnancy test is negative.
* Ability of reading, comprehending and finishing trial questionnaires and record, including VAS (Visual Analogue Scale) question.
* Before subject registration, written informed consent must be given according to local regulations.

Exclusion Criteria:

* Pregnant women without morning sickness.
* Presence of gastrointestinal tract obstruction or electrolyte imbalance.
* Any history of central nervous system disease(e.g. Primary brain tumour, seizure not controlled with standard medical therapy, brain metastases or history of stroke).
* Contraindication of glucocorticoid:1.Infection of virus, bacteria or fungus uncontrolled by antibiotics; 2.Active stomach or duodenum ulcer; 3.Severe hypertension, atherosclerosis, diabetes; 4.Osteoporosis;5.Corneal ulcer; 6.Pregnancy; 7.Reparative phase of trauma, operation or fraction; 8.Hypercortisolism; 9.Severe mental disorder or epilepsy; 10.Inadequate cardiac or renal function.
* Mental disability or severe emotional or mental disorder.
* Active infection(e.g. pneumonia, hepatitis) or any uncontrolled disease(e.g.diabetic ketoacidosis) that may affect study outcome or expose patients to unnecessary risk.
* Usage of any illicit drug, including medical marijuana or alcohol abusing(China drug dependence criteria).
* Treatment of unapproved medicine in the previous 4 weeks.
* Concomitant therapy of psychotropic medicine such as olanzapine.
* Hypersensitivity history towards Aprepitant, 5-HT3 receptor antagonist or dexamethasone.
* Previous treatment of Aprepitant.
* Unable to swallow capsules.
* Main researchers considered that the patient is unsuited to the trial.
* Unable or unwilling to follow research programme.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 248 (Actual)
Dates: Start 2015-08-04 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Complete response rate during the overall phase | Up to 1-2 months
  The proportion of patients without emesis episodes or rescue medication use during the overall phase (0-120 h)

SECONDARY OUTCOMES:
Complete response rate in the acute phase | Up to 1-2 months
  The proportion of patients without emesis episodes or rescue medication use during the acute phase (0-24h)
Complete response rate in the delayed phase | Up to 1-2 months
  The proportion of patients without emesis episodes or rescue medication use during the delayed phase (25-120 h)
No vomiting rate in the acute phase, delayed phase and overall phase | Up to 1-2 months
  The proportion of no vomiting (no vomiting or retching episodes) in the acute phase, delayed phase and overall phase
Affection caused by CINV reported by patients | Up to 1-2 months
Effects of CINV on daily life | Up to 1-2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Wang DS, Hu MT, Wang ZQ, Ren C, Qiu MZ, Luo HY, Jin Y, Fong WP, Wang SB, Peng JW, Zou QF, Tan Q, Wang FH, Li YH. Effect of Aprepitant for the Prevention of Chemotherapy-Induced Nausea and Vomiting in Women: A Randomized Clinical Trial. JAMA Netw Open. 2021 Apr 1;4(4):e215250. doi: 10.1001/jamanetworkopen.2021.5250. PMID 33835174